CLINICAL TRIAL: NCT05816330
Title: Safety and Efficacy of L9LS, a Human Monoclonal Antibody Against Plasmodium Falciparum, in a Randomized, Double-Blind, Placebo-Controlled Trial of Adults in Mali
Brief Title: L9LS MAb in Malian Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); Malaria Research and Training Center, Bamako, Mali (Other); University of the Sciences, Techniques and Technologies of Bamako (Other); University of Washington (Other); Harvard School of Public Health (HSPH) (Other); Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023/109/CE/USTTB
Record Dates: First submitted 2023-03-31; First posted 2023-04-18 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Plasmodium Falciparum Infection; Malaria
Keywords: Malaria; Plasmodium falciparum; L9LS; Monoclonal antibodies
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- L9LS 900 mg (Experimental): Adult participants receive a single dose of L9LS 900 mg subcutaneously.
  Interventions: Biological: L9LS (VRC-MALMAB0114-00-AB)
- Placebo (Placebo Comparator): Adult participants receive a single dose of Placebo subcutaneously.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: L9LS (VRC-MALMAB0114-00-AB) — Administered one time via subcutaneous route.
  Arms: L9LS 900 mg
Other: Placebo — Normal saline administered one time via subcutaneous route.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of a one time SC administration of L9LS in healthy adults in Mali, as well as its protective efficacy against naturally occurring Plasmodium falciparum (Pf) infection over a 6-month malaria season. A secondary objective is to determine if SC administration of L9LS at 900 mg (compared to placebo) mediates protection against naturally occurring Pf infection in healthy Malian adult females stratified by weight during a single malaria season.

DETAILED DESCRIPTION:
A phase 2 trial evaluating the safety and tolerability of a one time subcutaneous (SC) administration of L9LS, as well its protective efficacy against naturally occurring Pf infection over a 6-month malaria season. The primary study hypotheses is that L9LS will be safe and protective against malaria infection. As a secondary objective, the efficacy of L9LS within three body weight strata among female participants will each be compared to placebo. Before study agent administration, all subjects will be given artemether lumefantrine to clear any preexisting Pf blood stage infection.

The study is a randomized, double-blind, placebo-controlled, sex-stratified (2:1 female to male ratio) and weight-stratified trial (N=288 total) with 2 treatment arms: L9LS 900 mg SC (n=216) and placebo (n=72) to assess safety and protective efficacy of L9LS compared to placebo.

Subjects will receive the study agent and be followed at study visits 1, 3, 7, 14, 21, and 28 days later, and once every 2 weeks thereafter through 24 weeks. Primary study assessments include physical examination and blood collection for identification of Pf infection and other research laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged ≥18 and ≤49 years and weighing ≥ 45.0 and ≤ 90.0 kg.
2. Males aged ≥18 and ≤55 years and weighing ≥ 50.0 and ≤ 100.0 kg.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. In good general health and without clinically significant medical history.
5. Able to provide informed consent.
6. Willing to have blood samples and data stored for future research.
7. Resides in or near Kalifabougou, Faladje, or Torodo, Mali, and available for the duration of the study.
8. Females of childbearing potential must be willing to use reliable contraception from 21 days prior to study day 0 through the final study visit as described below.

   1. Reliable methods of birth control include 1 of the following: confirmed pharmacologic contraceptives via parenteral delivery or intrauterine or implantable device.
   2. Nonchildbearing women will be required to report date of last menstrual period, history of surgical sterility (i.e., tubal ligation, hysterectomy) or premature ovarian insufficiency, and will have urine or serum pregnancy tests performed per protocol.

Exclusion Criteria:

1. Pregnancy, as determined by a positive urine or serum beta-human choriogonadotropin (β hCG) test (if female).
2. Currently breastfeeding.
3. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and comply with the study protocol.
4. Study comprehension examination score of <80% correct or per investigator discretion.
5. Hemoglobin, white blood cell, absolute neutrophil, or platelet count outside the local laboratory-defined limits of normal. (Subjects may be included at the investigator's discretion for "not clinically significant" values.)
6. Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal. (Subjects may be included at the investigator's discretion for "not clinically significant" values.)
7. Infected with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
8. Known or documented sickle cell disease by history. (Note: Known sickle cell trait is NOT exclusionary.)
9. Clinically significant abnormal electrocardiogram (ECG; QTc >460 or other significant abnormal findings, including unexplained tachycardia or bradycardia).
10. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
11. Receipt of any investigational product within the past 30 days.
12. Participation or planned participation in an interventional trial with an investigational product until the last required protocol visit. [Note: Past, current, or planned participation in observational studies is NOT exclusionary; participation in the placebo arm of the Mali adult CIS43LS MAb trial (ClinicalTrials.gov Identifier: NCT04329104) is NOT exclusionary.]
13. Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
14. History of a severe allergic reaction or anaphylaxis.
15. Severe asthma (defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years, or that has required the use of oral or parenteral corticosteroids at any time during the past 2 years).
16. Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjögren's syndrome, or autoimmune thrombocytopenia.
17. Salivary gland disorder diagnosed by a doctor (e.g., parotitis, sialadenitis, sialolithiasis, salivary gland tumors).
18. Known immunodeficiency syndrome.
19. Known asplenia or functional asplenia.
20. Use of chronic (≥14 days) oral or IV corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of day 0.
21. Receipt of a live vaccine within the past 4 weeks or a killed vaccine within the past 2 weeks prior to study agent administration.
22. Receipt of immunoglobulins and/or blood products within the past 6 months.
23. Previous receipt of an investigational malaria vaccine or monoclonal antibody in the last 5 years.
24. Known allergies or contraindication against artemether lumefantrine.
25. Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of a subject participating in the trial, interfere with the evaluation of the study objectives, or render the subject unable to comply with the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 490 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-02-11 (Actual); Study Completion 2024-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kassoum Kayentao, MD, MPH, PhD, Principal Investigator — Faculté de Médecine Pharmacie d'Odontostomatologie (FMPOS); Peter Crompton, MD, MPH, Principal Investigator — National Institutes of Health (NIH)
Locations (3):
- Mali (3):
  - Faladje MRTC Clinic, Faladiè, Koulikoro
  - Kalifabougou MRTC Clinic, Kalifabougou, Koulikoro
  - Torodo MRTC Clinic, Torodo, Koulikoro

IPD SHARING:
Plan to Share IPD: Yes
Human data generated in this study for future research will be shared as follows:
  * De-identified or identified data with approved outside collaborators under appropriate agreements.
  * De-identified results or data in publication and/or public presentations.
Supporting Information: Study Protocol
Time Frame: Data will be shared at the time of publication or shortly thereafter.
Access Criteria: Data from this study may be requested from other researchers indefinitely after the completion of the primary endpoint by contacting Laboratory of Immunogenetics at NIH

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 490 participants were consented:
  * 156 participants were screen failure and ineligible
  * 45 participants served as backup
  * One participant withdrew consent
  * 288 participants received intervention
Period: Overall Study
Arm/Group | L9LS 900 mg | Placebo
Started | 217 | 71
Completed | 213 | 70
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | L9LS 900 mg | Placebo | Total
Number analyzed (Participants) | 217 | 71 | 288
Age, Customized [Count of Participants; unit: Participants]
  18-20 years | 31 | 7 | 38
  21-30 years | 61 | 19 | 80
  31-40 years | 72 | 18 | 90
  41-49 years | 48 | 22 | 70
  50-55 years (Male only) | 5 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 22 | 96
  Male | 143 | 49 | 192
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 217 | 71 | 288
Region of Enrollment [Number; unit: participants]
  Mali | 217 | 71 | 288

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local Adverse Events (AEs)
Description: Number of participants with local adverse events occurring within 7 days after administration of L9LS. Local reactogenicity included pain/tenderness, swelling, redness, bruising, and pruritus at the site of infusion. Adverse events were captured by Investigator examination and history from participants.
Time Frame: Within 7 days after administration of intervention
Population: All participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | L9LS 900 mg | Placebo
Number analyzed (Participants) | 217 | 71
Participants
  Injection site swelling | 7 | 1
  Pain at Injection site | 0 | 0
  Tenderness at injection site | 0 | 0
  Redness at injection site | 0 | 0
  Bruising at injection site | 0 | 0
  Pruritus at injection site | 0 | 0

2. Primary Outcome: Number of Participants With Systemic Adverse Events (AEs)
Description: Number of participants with local adverse events occurring within 7 days after administration of L9LS. Systemic reactogenicity events included fever, feeling unusually tired or unwell, muscle aches, headache, chills, nausea, and joint pain. Adverse events were captured by Investigator examination and history from participants.
Time Frame: Within 7 days after administration of intervention
Population: All participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | L9LS 900 mg | Placebo
Number analyzed (Participants) | 217 | 71
Participants
  Fever | 1 | 0
  Malaise | 0 | 0
  Muscle aches | 0 | 0
  Headache | 21 | 4
  Chills | 0 | 2
  Nausea | 2 | 0
  Joint pain | 0 | 0

3. Primary Outcome: Number of Participants With Local Adverse Events (AEs) (by Grade)
Description: The severity of local AEs was graded using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Clinical Trials
  Grade 1: Pain = does not interfere with activity; Tenderness = mild discomfort to touch; Erythema/Redness = 2.5-5 cm; Induration/Swelling = 2.5-5 cm and does not interfere with activity.
  Grade 2: Pain = Repeated use of non-narcotic pain reliever > 24 hours or interferes with daily activity; Tenderness= Discomfort with movement; Erythema/Redness = 5.1-10 cm; Induration/Swelling = 5.1-10 cm and interferes with activity.
  Grade 3: Pain = Any use of narcotic pain reliever or prevents daily activity; Tenderness = Significant discomfort at rest; Erythema/Redness = > 10 cm; Induration/Swelling = > 10 cm or prevents daily activity.
  Grade 4: Pain = Emergency room (ER) visit or hospitalization; Tenderness = ER visit or hospitalization; Erythema/Redness = Necrosis or exfoliative dermatitis; induration/Swelling = Necrosis Grade 5: Death
Time Frame: Within 7 days after administration of intervention
Population: All participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | L9LS 900 mg | Placebo
Number analyzed (Participants) | 217 | 71
Participants
  Grade 1 | 7 | 1
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

4. Primary Outcome: Number of Participants With Systemic Adverse Events (AEs) (by Grade)
Description: The severity of systemic adverse events occurring after the administration of L9LS was assessed using the grading scale below:
  Grade 1: Fever = 37.5^oC-37.9^oC; Fatigue, Headache, Myalgia = No interference with activity; Nausea = no interference with activity or 1-2 episodes/hour
  Grade 2: Fever = 38^oC-38.4^oC; Fatigue, Myalgia = Some interference with activity; Headache = Repeated use of non-narcotic pain reliever > 24 hours or some interference with activity; Nausea = Some interference with activity or > 2 episodes/24 hours
  Grade 3: Fever = 38.5^oC-39.5^oC; Fatigue = Prevents daily activity; Headache =Significant; any use of narcotic pain reliever or prevents daily activity; Myalgia =Significant; prevents daily activity; Nausea = Prevents daily activity, requires outpatient intravenous hydration
  Grade 4: Fever = > 39.5^oC; Fatigue, Headache, Myalgia = Emergency room (ER) visit or hospitalization; Nausea = ER visit or hospitalization for hypotensive shock
  Grade 5: Death
Time Frame: Within 7 days after administration of intervention
Population: All participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | L9LS 900 mg | Placebo
Number analyzed (Participants) | 217 | 71
Participants
  Grade 1 | 11 | 2
  Grade 2 | 13 | 4
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

5. Primary Outcome: Participants With Plasmodium Falciparum (Pf) Infection Detected by Microscopic Examination for Thick Blood Smear
Description: Number of participants with Plasmodium falciparum (Pf) blood stage infection defined as blood smear-positive for Pf was assessed by microscopic examination of thick blood smear collected from participants from day 7 through week 24 (168 days) after administration of L9LS or placebo. Sample was collected every two weeks from day seven until week 24. Analysis was done as number of participants who had at least one positive blood smear.
Time Frame: Day 7 through week 24
Population: All participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | L9LS 900 mg | Placebo
Number analyzed (Participants) | 217 | 71
Participants | 33 | 40

6. Secondary Outcome: Participants With Plasmodium Falciparum (Pf) Infection Detected by Real-Time Polymerase Chain Reaction (RT-PCR)
Description: Number of participants with Plasmodium falciparum (Pf) blood stage infection defined as blood sample positive for Pf was assessed by real-time polymerase chain reaction (RT-PCR) of blood sample collected from participants from day 7 through week 24 (168 days) after administration of L9LS or placebo. Sample was collected every two weeks from day seven until week 24. Analysis was done as number of participants who had at least one positive blood sample.
Time Frame: Day 7 through week 24
Population: All participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | L9LS 900 mg | Placebo
Number analyzed (Participants) | 217 | 71
Participants | 68 | 43

7. Secondary Outcome: Maximum Total Plasma Concentration (Cmax) for L9LS
Description: Maximum total plasma concentration (Cmax) following a 900 mg dose of L9LS. Serum collected on days 0, 1, 7, 14, 28, 56, 84, 112, 140, & 168 after the administration of L9LS. Cmax for L9LS was obtained directly by visual inspection of the plasma concentration versus time profiles postdose. Analysis was done to determine each participant's observed maximum concentration based on all available timepoints and cumulative output was calculated as the central tendency and dispersion metric based on the observed maximum concentrations.
Time Frame: Measure through week 24
Population: Per protocol document, measure apply to participants who received L9LS
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | L9LS 900 mg
Number analyzed (Participants) | 217
ug/mL | 158.07 (30.41)

8. Secondary Outcome: Time to Maximum Plasma Concentration (TMax) for L9LS - Hours
Description: Time to maximum total plasma concentration (Cmax) following a 900 mg dose of L9LS on day 7 post administration of drug. Tmax for L9LS was obtained directly by visual inspection of the plasma concentration versus time profiles. Analysis was done to determine the time (in hours) at which the maximum observed concentration was achieved for each participant and cumulative output was calculated as the central tendency and dispersion metric based on the observed time of maximum concentration.
Time Frame: Day 7 post administration of drug
Population: Per protocol document, measure apply to participants who received L9LS.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | L9LS 900 mg
Number analyzed (Participants) | 217
Hours | 172.9 (30.0)

9. Secondary Outcome: Time to Maximum Plasma Concentration (TMax) for L9LS - Days
Description: Time to maximum total plasma concentration (Cmax) following a 900 mg dose of L9LS. Serum collected on days 0, 1, 7, 14, 28, 56, 84, 112, 140, & 168 after the administration of L9LS. Tmax for L9LS was obtained directly by visual inspection of the plasma concentration versus time profiles. Analysis was done to determine the time (in days) at which the maximum observed concentration was achieved for each participant and cumulative output was calculated as the central tendency and dispersion metric based on the observed time of maximum concentration.
Time Frame: Measure through week 24
Population: Per protocol document, measure apply to participants who received L9LS.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | L9LS 900 mg
Number analyzed (Participants) | 217
Days | 7.20 (1.25)

ADVERSE EVENTS:
Time Frame: Up to 24 weeks from administration of intervention
Arm/Group | L9LS 900 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/217 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/217 | 1/71
Other Adverse Events (participants affected / at risk) | 192/217 | 57/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L9LS 900 mg (N=217) | Placebo (N=71)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L9LS 900 mg (N=217) | Placebo (N=71)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 21 (21) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Bradycardia (Cardiac disorders) | 4 (4) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 4 (6)
Dental Caries (Gastrointestinal disorders) | 11 (12) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 32 (39) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 2 (2)
Toothache (Gastrointestinal disorders) | 24 (26) | 3 (3)
Vomiting (Gastrointestinal disorders) | 8 (9) | 5 (5)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (2) | 0 (0)
Chills (General disorders) | 15 (16) | 5 (5)
Injection Site Swelling (General disorders) | 7 (7) | 1 (1)
Pyrexia (General disorders) | 10 (10) | 2 (2)
Conjunctivitis (Infections and infestations) | 17 (18) | 6 (6)
Dysentery (Infections and infestations) | 2 (2) | 3 (3)
Furuncle (Infections and infestations) | 4 (4) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Genital Infection (Infections and infestations) | 6 (6) | 1 (1)
Genitourinary Tract Infection (Infections and infestations) | 4 (4) | 2 (2)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 20 (20) | 23 (26)
Mastitis (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 3 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 3 (3)
Rhinitis (Infections and infestations) | 42 (49) | 17 (24)
Salmonellosis (Infections and infestations) | 3 (3) | 1 (1)
Tinea Infection (Infections and infestations) | 1 (1) | 0 (0)
Tinea Pedis (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 37 (39) | 14 (14)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 1 (1) | 0 (0)
Blood Pressure Diastolic Decreased (Investigations) | 1 (1) | 0 (0)
Blood Pressure Diastolic Increased (Investigations) | 2 (2) | 0 (0)
Blood Pressure Increased (Investigations) | 1 (3) | 0 (0)
Blood Pressure Systolic Increased (Investigations) | 2 (2) | 1 (1)
Haemoglobin Decreased (Investigations) | 1 (1) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 4 (4)
Headache (Nervous system disorders) | 112 (167) | 24 (38)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (31) | 8 (10)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Tooth Extraction (Surgical and medical procedures) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT05816330/Prot_SAP_000.pdf